CLINICAL TRIAL: NCT06787313
Title: Precision Palliative Care for Patients With Advanced Esophageal Cancer: a Randomized Phase III Trial
Brief Title: Precision Palliative Care for Patients With Advanced Esophageal Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Prof., Fudan University
Other Study IDs: ESO-Shanghai25
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer
Keywords: Precision palliative Care; immunotherapy; PD-1
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Arm: All participants receive standard oncologic palliative care.
- Supportive Arm: All participants receive precision palliative care based on scale screening result.
  Interventions: Other: precision palliative care

INTERVENTIONS:
Other: precision palliative care — Participants receive precision palliative care based on scale screening result.
  Groups: Supportive Arm

SUMMARY:
The goal of this clinical trial is to learn if precision palliative care improves survival of patients with advanced esophageal cancer in adults.

Researchers will compare precision palliative care and standard palliative care to see if precision palliative care works more effectively to treat advanced esophageal s cancer.

Participants will receive precision palliative care or standard palliative care. All participants will answer survey questions about their quality of life, MDASI, PHQ-9, GAD-7 for 1 years.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged ≥18 years
3. Histologically confirmed esophageal cancer
4. Clinical stages IV based on the 8th AJCC TNM classification, or recurrent esophageal cancer
5. plan to treated with anti-PD-1/PD-L1 immunotherapy
6. Eastern Cooperative Oncology Group(ECOG) performance status: 0-2
7. Adequate organ functions Absolute neutrophil counts (ANC) ≥1.5×109⁄L; Hemoglobin (Hb) ≥9g⁄dl; Platelet (Plt) ≥100×109⁄L; Total bilirubin ≤1.5 upper limit of normal (ULN); Aspartate transaminase (AST) ≤2.5 ULN; Alanine aminotransferase (ALT) ≤2.5 ULN; Creatinine ≤1.5 ULN.

Exclusion Criteria:

1. Esophageal perforation or hematemesis
2. Any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism and hypothyroidism (effective hormone replacement therapy excepted)) and immunosuppressive agents or systemic hormonal therapy indicated within 28 days (for adverse events of chemoradiotherapy excepted).
3. Disease progression occurs within 3months after anti-PD-1/PD-L1 immunotherapy.
4. Allergic to macromolecular protein preparations, or to any of the ingredients in anti-PD-1/PD-L1 inhibitors for injection.
5. Uncontrolled heart diseases or clinical symptoms, such as: (1) New York Heart Association(NYHA) class II or higher heart failure; (2) unstable angina; (3) myocardial infarction within 1 year; (4)clinically significant arrhythmia requiring clinical intervention.
6. Congenital or acquired immunodeficiency (such as HIV infection); active hepatitis B (HBV-DNA≥104 copy number/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method); active tuberculosis.
7. Active infection or unexplained fever >38.5 °C within 2 weeks before randomization (fever due to tumor excepted, according to investigator).

   Patients with fertility reluctant to take contraceptive measures during the trial, or female patients pregnant or breastfeeding.
8. According to the investigator, other factors that may cause termination of the study. ie, other serious diseases (including mental illness) require combined treatment, family or social factors, which may affect the safety or the collection of trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in this study, all subjects are diagnosed with stages IV esophageal cancer or recurrent esophageal cancer. All subjects plan to treated with anti-PD-1/PD-L1 immunotherapy. Subjects are inpatients or outpatients.
Sampling Method: Probability Sample
Enrollment: 624 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival for all patients

SECONDARY OUTCOMES:
Quality of life | 1 year
  Quality of life for all patients
PFS | 2 years
  PFS for all patients
biomarker | 2 years
  biomarker to predict immunotherapy effect

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided